CLINICAL TRIAL: NCT03480516
Title: Efficacy of Silver Diamine Fluoride (SDF) and Fluoride Varnish in Arresting and Preventing Dental Caries in Primary School Children: Randomized Controlled Clinical Trial
Brief Title: Comparison of Caries Arrested & Prevented Among SDF, NaF Varnish and Combination in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Kemporn Kitsahawong, Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KKUHE602106
Record Dates: First submitted 2018-03-11; First posted 2018-03-29 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2018-09

CONDITIONS: Dental Caries in Children; Satisfaction; Cost Effectiveness; Oral Health; Quality of Life
Keywords: Silver Diamine Fluoride; Sodium Fluoride Varnish; Arrest caries; Caries prevention; Cost Effectiveness; Oral Health; Quality of Life
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SDF arm (Experimental): SDF arm is application of 38% silver diamine fluoride solution (SDF) on cavitated caries in primary molar, , cavities in anterior teeth will be applied only on additional consent obtained.
  Interventions: Device: SDF
- Fluoride varnish arm (Experimental): Fluoride varnish arm is application of 5% sodium fluoride varnish on all surface of every tooth.
  Interventions: Device: Fluoride varnish
- Combination arm (Experimental): Combination arm is application of 38% silver diamine fluoride solution(SDF) on cavitated caries in primary molar, , cavities in anterior teeth will be applied only on additional consent obtained and then apply of 5% sodium fluoride varnish on all surface of every tooth.
  Interventions: Device: SDF; Device: Fluoride varnish

INTERVENTIONS:
Device: SDF — 38% silver diamine fluoride solution
  Other Names: Silver diamine fluoride
  Arms: Combination arm; SDF arm
Device: Fluoride varnish — 5% sodium fluoride varnish
  Other Names: Sodium fluoride varnish
  Arms: Combination arm; Fluoride varnish arm

SUMMARY:
Tooth decay is one of the most common chronic infectious disease found in children worldwide and if left untreated, is rapidly progress. Severe tooth decay in children is not only affect child's health and school performance, but also has impact on the family well-being. Oral rehabilitation in children requires time, resources and effort of dental specialists, the child and parents. Caries is a destructive condition of organic and inorganic components of the tooth structures but reversible and most importantly, preventable. Topical fluoride therapy, delivered by dentists has been effectively used to speed up the repair process as well as to strengthen the surface of intact tooth structure. Topical fluoride is available in various preparations. Regular application of sodium fluoride varnish is every three months, by far, considered as effective method in preventing new caries, particularly in the high-risk children. It has the advantage of containing therapeutic concentration of fluoride and ability to flow over and stick to the tooth surface. Whereas silver ion and relatively higher fluoride concentration in Silver Diamine Fluoride (SDF) has been shown to be the most effective in harden the decay, stop the caries progress and eliminate pathogenic bacteria. It can be hypothesize that when use in combination in school children, both reagents might have synergistic effect on arresting existing caries as well as preventing new caries.

DETAILED DESCRIPTION:
Fluoride varnish is a good choice to consider. For caries prevention in young children, It has high efficacy in caries prevention.

Fluoride varnish has a high F concentration and prolong contact time with enamel, So it can prevent new caries and remineralize initial enamel caries. Silver diamine fluoride solution is effective in arresting dentine caries. Silver diamine fluoride has high fluoride concentration and contain silver ion. when apply dentine caries or cavitated caries can increase hardness of dentine and arresting caries.

When use in combination, it might enhance, the Efficacy in Arresting and Preventing Dental Caries in children

ELIGIBILITY:
Inclusion Criteria:

* School children aged 6- 7 years old.
* Have at least one or more active dentin caries lesions in primary canine/molar.
* Parents give consent.

Exclusion Criteria:

* Uncooperative child
* Allergic reaction to silver or materials containing adhesive.
* Received topical fluoride 3 months prior to enrollment.
* Primary carers are unable to response to questionnaire.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Number of arrested caries lesion changed from baseline | 18 months
  Number of arrested caries lesion changed from baseline. The arresting dentine caries lesion was evaluated at 18 months after first application. Evaluation criteria included the condition of the hardness and discoloration of carious lesion. The carious lesion was re-categorized as a binary outcome: Dental caries (active/inactive)

SECONDARY OUTCOMES:
Increasing number of new caries lesion from baseline | 6 months
  The dental caries status was evaluated at 6 months after fluoride application. Evaluation criteria included decay(d), missing(m), filling(f) index
Increasing number of new caries lesion from baseline | 12 months
  The dental caries status was evaluated at 12 months after fluoride application. Evaluation criteria included decay(d), missing(m), filling(f) index
Increasing number of new caries lesion from baseline | 18 months
  The dental caries status was evaluated at 18 months after fluoride application. Evaluation criteria included decay(d), missing(m), filling(f) index
Parental satisfaction | 2 weeks
  parental satisfaction will be collected, by a seft-administered questionnaire, at 2 weeks.
Parental satisfaction | 18 months
  parental satisfaction will be collected, by a seft-administered questionnaire, at 18 months
Child satisfaction | 6 months
  Child satisfaction will be collected after fluoride application by interview. at 6 months
Child satisfaction | 12 months
  Child satisfaction will be collected after fluoride application by interview. at 12 months
Child satisfaction | 18 months
  Child satisfaction will be collected after fluoride application by interview. at 18 months
Cost Effectiveness | 18 months
  Cost effectiveness analysis of arrested caries lesion and new caries lesion at 18 months
Oral Health-Related Quality of life | 12 months
  Oral health related quality of life in children is being measured using the Child-Oral Impacts on Daily Performance Index (Child-OIDP) at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kemporn Kitsahawong, DDS., MSc., Principal Investigator — Faculty of Dentistry, Khon Kaen University
Locations (1):
- Faculty of Dentistry , Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No